CLINICAL TRIAL: NCT05034601
Title: Comparison of Erector Spinae Plane and Paravertebral Nerve Blocks for Postoperative Analgesia in Children After the Nuss Procedure
Brief Title: ESPB vs TPVB for Postoperative Analgesia After the Nuss Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Min Xu, Department of Anesthesiology, West China Hospital, Sichuan University, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2021-866
Record Dates: First submitted 2021-08-21; First posted 2021-09-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Nerve Block; Analgesia; Pectus Excavatum
MeSH Terms: conditions — Agnosia; Funnel Chest

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB group (Experimental): 0.25% ropivacaine 0.5 ml/kg is injected at the fascial plane deep to the erector spinae muscle
  Interventions: Procedure: ESPB group
- TPVB group (Active Comparator): 0.25% ropivacaine 0.5 ml/kg is injected into the thoracic paravertebral space (T5) using TPVB approach.
  Interventions: Procedure: TPVB group

INTERVENTIONS:
Procedure: ESPB group — A 21-gauge 100-mm needle will be inserted into the fascial layer beneath the iliocostalis, longissimus, and spinalis muscles. A bolus of 0.25% ropivacaine 0.5 ml/kg will be injected into the fascial layer. Contralateral ESPB will be performed similarly.
  Other Names: Erector spinae plane block
  Arms: ESPB group
Procedure: TPVB group — A 21-gauge 100-mm insulated needle will be inserted into the paravertebral space via an in-plane parasagittal approach. After perforating the costotransverse ligament, 0.25% ropivacaine 0.5 ml/kg will be injected. Anterior movement of the pleura indicated the appropriate spread of the local anesthetics in the paravertebral space. The process will be repeated on the contralateral side.
  Other Names: Thoracic paravertebral block
  Arms: TPVB group

SUMMARY:
This is a prospective randomized double-blind non-inferiority trial designed to test the hypothesis that erector spinae plane block (ESPB) is non-inferior to thoracic paravertebral block (TPVB) in postoperative pain control after pectus excavatum repair.

ELIGIBILITY:
Inclusion Criteria:

* Age between 4 to 18 years Scheduled for elective Nuss surgery Written informed consent is obtained from parents of each patient.

Exclusion Criteria:

* Coagulation dysfunction. American Society of Anesthesiologists Physical Status 4 or 5. Allergy to study medication. Local infection at the site of injection or systemic infection. Inability to understand Chinese.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Pain scores at rest at 24 hours postoperatively | 24 hours postoperatively
  Pain scores will be recorded using the Numeric Rating Scale (NRS) scores (0-10).

SECONDARY OUTCOMES:
The pain degree at rest and after movement or coughing(dynamic) | at 3, 6, 12, 24, and 48 hours after surgery
  The pain degree at rest and after movement or coughing at 3, 6, 12, 24, and 48 hours after surgery respectively.
total rescue morphine-equivalent consumption per weight | at 24 and 48 hours after surgery
  total rescue morphine-equivalent consumption per weight at predetermined time intervals (24 and 48 hours) after surgery
Emergence agitation at 5, 15, 30 min after extubation | at 5, 15, 30 min after extubation
  Emergence agitation will be registered using pediatric anesthesia emergence delirium (PAED) at 5, 15, 30 min after extubation
Total dosage of intraoperative sufentanil and remifentanil | during surgery
  Total dosage of intraoperative sufentanil and remifentanil per weight
The time to first analgesia request | within the 3 days after surgery
  Time from operation to first rescue analgesia request
The time to first mobilization | within the 3 days after surgery
  Time from operation to ambulation
Side effects | within the 5 days after surgery
  Side effects such as pneumothorax, local anesthetic toxicity, postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Jin Liu, Study Chair — Department of Anesthesiology, West China Hospital, Sichuan University
Locations (1):
- Department of Anesthesiology, West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu M, Zhang G, Gong J, Yang J. Comparison of erector spinae plane and paravertebral nerve blocks for postoperative analgesia in children after the Nuss procedure: study protocol for a randomized controlled non-inferiority clinical trial. Trials. 2022 Feb 14;23(1):139. doi: 10.1186/s13063-022-06044-y. PMID 35164831